CLINICAL TRIAL: NCT06981923
Title: Awake Bedside Assessment of The Airway and Evaluation of Tracheal Intubation With CMAC D-Blade or Video Stylet in Bariatric Surgery: A Randomized Comparative Study
Brief Title: Awake Bedside Assessment of The Airway and Evaluation of Tracheal Intubation With CMAC D-Blade or Video Stylet in Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Responsible Party: Principal Investigator, Mohamed Hany Ashour, Professor of General surgery, Surgeon, General Committee of Teaching Hospitals and Institutes, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CMAC D-Blade or Video Stylet
Record Dates: First submitted 2025-05-11; First posted 2025-05-21 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Difficult Intubation in Obesity
Keywords: CMAC D-Blade; CMAC Video-style; bariatric patients; Simplified Airway Risk Index (SARI)

STUDY DESIGN:
Intervention Model Description: Intervention Groups
  1. CMAC D-Blade Group: Intubation will be performed using the CMAC D-Blade.
  2. CMAC Video Style Group: Intubation will be performed using the CMAC Video stylet.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CMAC D-Blade Group (Active Comparator): Intubation will be performed using the CMAC D-Blade
  Interventions: Device: CMAC D-Blade
- CMAC Video Style Group (Active Comparator): Intubation will be performed using the CMAC Video stylet
  Interventions: Device: CMAC Video Stylet

INTERVENTIONS:
Device: CMAC D-Blade — Intubation will be performed using the CMAC D-Blade
  Arms: CMAC D-Blade Group
Device: CMAC Video Stylet — Intubation will be performed using the CMAC Video stylet
  Arms: CMAC Video Style Group

SUMMARY:
Patients undergoing bariatric surgery often present challenges during intubation due to limited neck mobility, increased soft tissue in the airway, and elevated body mass index (BMI). Predicting difficult intubation in these patients is critical to ensuring safety. The Simplified Airway Risk Index (SARI) by Ganzouri is a validated tool for predicting difficult intubation. It considers factors like neck mobility, Mallampati score, and body weight, which are highly relevant in difficult airway prediction in the bariatric population.

The CMAC video laryngoscope is widely used to manage difficult airways. Two commonly used devices are the CMAC D-Blade, designed explicitly for difficult airways, and the CMAC Video stylet, which combines video guidance with a flexible tip. This study will compare the efficacy and safety of these two devices in bariatric patients with an anticipated difficult airway, as identified by the SARI.

DETAILED DESCRIPTION:
Comparing the effectiveness and safety of the CMAC D-Blade versus the CMAC Video-style for awake bedside airway assessment and their performance during tracheal intubation in bariatric patients with expected difficult intubation as predicted by the Simplified Airway Risk Index (SARI).

Standard monitoring will be attached and recorded. Preoperative awake airway assessment: after airway topicalization, both devices will be used for airway assessment according to the group allocation, and the Cormack and Leane will be recorded.

Induction of Anesthesia: A standardized protocol will be followed for all patients, including preoxygenation and administration of propofol, fentanyl, and muscle relaxants (e.g., rocuronium).

Intubation: The intubating anesthetist will use the assigned device.

- Rescue Strategy: If intubation fails after three attempts or exceeds 120 seconds, the anesthetist will switch to an alternative device or follow the institutional difficult airway protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years)
* BMI ≥ 35 kg/m²
* SARI score ≥ 4
* Scheduled for elective bariatric surgery

Exclusion Criteria:

1. SARI score < 4.
2. any known or suspected airway pathology (such as tumors, airway trauma, or history of airway surgery/tracheostomy).
3. Emergency surgery.
4. Coagulopathy.
5. seizures, pregnancy,
6. mouth opening ≤ 2 cm.
7. contraindications to general anesthesia or neuromuscular blockade and uncooperative patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2025-05-10 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
First-Pass Success Rate | At the time of the procedure
  This is a successful intubation on the first attempt without needing an alternative device.

SECONDARY OUTCOMES:
Time to Intubation | At the time of the procedure
  Measured from the insertion of the device into the mouth until confirmation of endotracheal tube placement via capnography.
Intubation Difficulty Score (IDS) | At the time of the procedure
  A composite score based on multiple intubation-related factors, such as the number of attempts, additional maneuvers, and the application of external laryngeal pressure.
Stress response of intubation | At the time of the procedure
  serum level of stress markers measured before and after intubation (catecholamines)
awake Cormack-Lehane Classification | At the time of the procedure
  awake Cormack-Lehane Classification of Glottic View assessment and after induction of anesthesia during the intubation process.
Operator satisfaction | At the time of the procedure
  the anesthesiologist rated their satisfaction with the device performance on a 5-point Likert scale (5 = extremely satisfied, 4 = satisfied, 3 = neutral, 2 = dissatisfied, 1 = extremely dissatisfied).
Complications | At the time of the procedure
  for example,
  1. Hypoxemia (SpO₂ < 92%)
  2. Esophageal intubation or failed intubation
  3. Airway trauma (dental or oropharyngeal injury)
Need for Alternative Intubation Devices | At the time of the procedure
  Documentation of cases where the initially assigned device failed, and an alternative was needed.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Madina Women's Hospital, Alexandria
  - The surgical department of Medical Research Institute Hospital, Alexandria University, Alexandria

IPD SHARING:
Plan to Share IPD: Yes
The analysis will be performed on a blinded dataset after completing the medical/scientific review. All protocol violations will be identified and resolved, and the dataset will be declared complete. All data will be collected in a data management system (Castor EDC, Amsterdam, The Netherlands; https://www.castoredc.com), handled according to Good Clinical Practice guidelines, Data Protection Directive certificate, and complied with Title 21 CFR Part 11. Furthermore, the data centers where all the research data will be stored are certified according to ISO27001, ISO9001, and Dutch NEN7510.
  Can be asked by the contact person
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Whole study period
Access Criteria: Ask contact person